CLINICAL TRIAL: NCT02632994
Title: Master Rollover Protocol for Continued Safety Assessment of Study Drug
Status: Available | Type: Expanded Access
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 16161; I8I-MC-JYAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — LY3023414

INTERVENTIONS:
Drug: LY2503029 — Administered orally.
Drug: LY3023414 — Administered orally.
Drug: LY3838915 — Administered orally.
Drug: LY3847429 — Administered orally.

SUMMARY:
This study is for patients who have participated in a previous study and who continue to receive benefit to have continued access to study drug and/or treatment.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible patients must be currently receiving benefit in a concluded Lilly study for a compound that has opened an addendum in the continued access protocol.

Exclusion Criteria:

* Patients must not be concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - UCLA Medical Center, Torrance, California
  - Fort Wayne Oncology & Hematology, Fort Wayne, Indiana
  - Sarah Cannon Cancer Center, Nashville, Tennessee